CLINICAL TRIAL: NCT06168669
Title: A Safety and Effectiveness Prospective Blinded Clinical Study to Validate xBar System as Monitoring Tool for Anastomotic Leaks Detection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Exero Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP03
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Surgery; Anastomotic Leak
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: All eligible subjects will be assigned with the investigational device.
Masking Description: Investigators, clinical teams and subjects will be blinded to the outcomes provided by xBar system. Post operative monitoring will be as per SOC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Singel arm (Other): All patients will be treated with the investigational device.
  Interventions: Diagnostic Test: xBar system

INTERVENTIONS:
Diagnostic Test: xBar system — xBar system is surgical drain with embedded sensors. Collected data will be evaluated for an ability to identify anastomotic leaks. The xBar system does not have therapeutic indication.

SUMMARY:
Purpose: To validate the safety and effectiveness of xBar monitoring tool for detection of post-operative anastomotic leaks in subjects undergoing rectal/sigmoid resections with anastomosis.

The clinical team is blinded to the leak detection of the xBar system.

DETAILED DESCRIPTION:
Study design: Pivotal, Prospective, Blinded, multi-center study. Study Population: This study will enroll approximately 190 eligible subjects undergoing scheduled colorectal surgery with anastomosis, without concomitant diversion.

xBar is an investigational device intended for post-op monitoring of patients undergoing GI surgery. The device is comprised of a surgical drain with embedded electrodes, connected to a small electronic device that records and relays data from the electrodes. The collected data is processed for early detection of complications.

Study description: The study is intended to validate the performance of the xBar system's anastomotic leak detection monitoring tool following colorectal resection with drain placement. During the index surgery the xBar device will be placed according to institution standard procedures and data recording will commence for a period of at least 3 days. Safety and complication detection performance will be evaluated retrospectively by comparing the diagnosis on a subject level done by the clinical team, who is blinded to xBar results, and the system.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 22 years
2. Indication for sigmoid or rectal resection surgery.
3. Usage of drain during the surgery (to be confirmed during the surgery)
4. Willing and able to comply with the study follow up.
5. Able and agree to provide an informed consent.

Exclusion Criteria:

1. Contraindication for surgery and/or general anesthesia.
2. Pregnancy or lactation.
3. Planned or unplanned fecal diversion during the surgery (to be confirmed during the surgery)
4. Known electronic device implanted in the chest or the abdominal cavity (e.g., pacemaker, cardioverter/defibrillator).
5. Major medical or psychiatric illness or condition, or other factors that may affect general health or ability to adhere to the follow-up schedule.
6. Known allergic reactions to materials used in the components of the xBar system, i.e., silicone, rubber and stainless-steel.
7. Participation in another interventional study during the xBar system usage.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-03-11 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety | through study completion, an average of 1 year
  Lack of unanticipated serious adverse events related to the xBar system or xBar procedure during the study period.
Safety - Severe leak rate - comparable to SOC. | through study completion, an average of 1 year
  Statistical evaluation of prevalence of anastomotic leaks in the study group compared to the prevalence present in the literature.
Performance - successful xBar placement. | through study completion, an average of 1 year
  The device is working properly and records data in 90% of the cases or more.
Performance - Sensitivity and Specificity of severe leak detection | through study completion, an average of 1 year
  Sensitivity and Specificity are non-inferior compared to Standard of care at POD 3

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Tampa, Tampa, Florida
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health, Detroit, Michigan
  - Bryan Medical Center, Lincoln, Nebraska
  - Weill Cornell MC, NY, New York, New York
  - Mount Sinai Health System, New York, New York
  - Northwell Health, NY, New York, New York
  - Stony Brook University Hospital and Cancer Center, New York, New York
  - HCA, Houston, Texas
- Israel (3):
  - Soroka MC, Beersheba
  - Rabin MC, Petah Tikva
  - Kaplan MC, Rehovot

IPD SHARING:
Plan to Share IPD: No